CLINICAL TRIAL: NCT04928235
Title: Utility of Thermal Imaging in Diagnosis of Cellulitis for Lower Extremity Complaints in the Emergency Department
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2018-0823 Phase 2; A534100 (Other: UW Madison); SMPH/EMERG MED (Other: UW Madison); 1K08HS024342-01A1 (AHRQ)
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Cellulitis; Skin and Subcutaneous Tissue Infection
Keywords: Diagnostic confidence; Diagnostic accuracy; Diagnostic error
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: All participants will have thermal imaging of their lower extremities. The temperature values will be shared with the attending physician. The physician will be asked questions about their diagnostic confidence before and after seeing the temperature values.
  Interventions: Diagnostic Test: Thermal Imaging as Diagnostic Adjunct

INTERVENTIONS:
Diagnostic Test: Thermal Imaging as Diagnostic Adjunct — Thermal images of the participants lower extremities will be taken and skin surface temperature values will be provided to the healthcare provider for review during the emergency department encounter.

SUMMARY:
The overall purpose of the study is to determine how providing physicians with a quantitative measure of skin surface temperature influences diagnoses and diagnostic confidence in potential cellulitis cases when added to the standard evaluation.

DETAILED DESCRIPTION:
Previous literature estimates the emergency department misdiagnosis rate for cellulitis exceeds 30% due to conditions which can mimic cellulitis (termed pseudocellulitis). These diagnostic errors are associated with an estimated $195 to $515 million dollars in avoidable healthcare spending each year. Objective skin surface temperature measurement, obtained via thermal imaging cameras, has been proposed as a diagnostic adjunct that may reduce diagnostic error in cases of suspected cellulitis. One recent study, identified that the maximum affected skin temperature in cellulitis is significantly higher than in pseudocellulitis, and the temperature gradient between affected and unaffected sites in patients with cellulitis is significantly higher than in patients with pseudocellulitis.

The overall purpose of the study is to determine how providing physicians with a quantifiable measure of skin surface temperature information influences diagnoses and diagnostic confidence in potential cellulitis cases when added to standard physical exam techniques

The Aims of the study are to :

Specific Aim 1: To characterize the temperature difference between affected and unaffected limbs in patients with cellulitis in the emergency department.

Specific Aim 2: To characterize the temperature difference between cases of cellulitis and pseudocellulitis

Specific Aim 3: To determine how quantifying temperature gradients changes diagnostic confidence and accuracy when added to the standard diagnostic evaluation for potential cellulitis.

The investigators will prospectively enroll a maximum of 560 patients with non-traumatic lower extremity dermatologic complaints with visible erythema (potential cellulitis) in the University of Wisconsin Emergency Department. A thermal image and a photograph of the affected and the unaffected limbs will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Participant is presenting to the University of Wisconsin Emergency Department
* Participant has an acute skin complaint on the lower extremity

Exclusion Criteria:

* Participant is has limited English and Spanish proficiency
* There was an acute traumatic injury of affected area in last 5 days- includes burns
* Affected area has a confirmed fracture
* Participant is pregnant
* Participant is a prisoner
* Current complaint is in an area of past surgical procedure (within past 4 weeks)
* Participant has implant or hardware at site
* Animal or human bite is cause of complaint
* Temperature of the leg has been altered in the last one hour
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Seeking to include all patients who present to the Emergency Department for a skin related, acute lower extremity complaint and able to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2021-07-18 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-02-18 (Actual)

PRIMARY OUTCOMES:
Skin Temperature Difference Between Affected and Unaffected Legs for Participants with Cellulitis | up to one hour
  Differences in skin surface temperatures of affected and unaffected areas for those with a final diagnosis of cellulitis.
Skin Temperature Difference Between Participants Diagnosed with Pseudocellulitis and Cellulitis | up to one hour
  Determine differences in skin surface temperatures between cases of pseudocellulitis and cellulitis (on the affected legs).

SECONDARY OUTCOMES:
Change in Diagnostic Confidence as Measured by Physician Self-Report | up to one hour
  Comparison of the change in diagnostic confidence as measured by the attending physician response pre/post thermal imaging review. This was a question developed by the study team and response options include not at all confident, slightly confident, somewhat confident, very confident, extremely confident. No number values are assigned to response values as of yet.
Diagnostic agreement with expert review panel | 6 months
  Provider cellulitis diagnostic assignment (yes/no) will be compared to an expert panel to determine the rate of concordance.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pulia, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Emergency Department, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No